CLINICAL TRIAL: NCT01034085
Title: Effects of Nicotine on Areas of Impaired and Preserved Functioning in Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909445; 09-DA-N445
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-06-11

CONDITIONS: Nicotine Dependence; Schizophrenia
Keywords: Nicotine; Schizophrenia; Cognition; Genes; Smoking; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Smoking; Cigarette Smoking

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Some people with schizophrenia have problems with their working memory and paying attention for extended periods. These difficulties cannot be treated with antipsychotic medications or with many standard therapies.
* The prevalence of cigarette smoking among individuals with schizophrenia is about three times higher than in the general population. Research has shown that nicotine, the addictive component found in cigarettes, can help improve attentional and working memory performance. Researchers are interested in learning more about whether there may be an overlap in the cognitive functions beneficially affected by nicotine and areas of dysfunction in individuals with schizophrenia.

Objectives:

* To evaluate the potential of transdermal nicotine to alleviate cognitive deficits in schizophrenia, and to determine whether naturally maintained cigarette-smoking, in comparison, is an effective self-medication.
* To gather preliminary data on genetics that may account for individual and group differences in the performance effects of nicotine.

Eligibility:

- Current smokers (25 or more cigarettes per week for at least 1 year) between 18 and 55 years of age who are either healthy volunteers or have been diagnosed with schizophrenia/schizoaffective disorder.

Design:

* The study will require five visits to the research center, with an initial screening visit, a training session, and three test sessions. Ideally, all visits will occur 1 week apart.
* Training session: Participants will receive training on the types of computerized cognitive and attentional behavior tests that will be given during the active portion of the study. Participants will also fill out questionnaires on nicotine use and other alcohol and drug use.
* Test sessions: Participants will be assigned to random groups and will complete tests that assess cognitive performance (a) while maintaining their usual smoking behavior, (b) after minimal deprivation (3.5 hours without smoking) while wearing a placebo patch, and (c) under the influence of a standard nicotine patch. The order of these sessions will be different for individual participants.
* Participants will provide blood samples throughout the research study for evaluation purposes.

DETAILED DESCRIPTION:
Objective:

1. To evaluate the potential of transdermal nicotine to alleviate distinct cognitive deficits in schizophrenia, and to determine whether naturally maintained cigarette-smoking, in comparison, is an effective self-medication.
2. To gather preliminary data on genotypes that may account for interindividual and group differences in the performance effects of nicotine.

Study population:

45 regular smokers with schizophrenia, 45 matched control smokers (greater than or equal to 5 cigarettes/day).

Design:

Double-blind, placebo-controlled, within-subject study, evaluating cognitive functions under conditions of normal smoking, transdermal nicotine (14 mg/day), and placebo (minimal tobacco deprivation).

Outcome measures:

Measures of cognitive task performance, measures of subjective state, plasma concentrations of nicotine and metabolites, and genotype with regards to genes coding for nicotinic receptor subunits, MAO, and COMT.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants:

1. Age 18 through 55. The aim is to minimize population inhomogeneity related to cognitive decline due to normal aging.
2. Smoker of 5 or more cigarettes, cigarillos or cigars per day, on 5 or more days/week, for at least the last 12 months
3. Normal or corrected to normal visual acuity (at least 20/100).

Participants with mental illness, additional inclusion criteria:

1. DSM-IV diagnosis of schizophrenia or schizoaffective disorder
2. Ability to give written informed consent
3. Four weeks of stable pharmacological treatment (same psychiatric medication at same dose)

EXCLUSION CRITERIA:

All participants:

1. History of myocardial infarction, heart failure, angina, stroke or severe arrhythmias, EKG abnormalities as specified under Screening methods
2. Uncontrolled high blood pressure (resting systolic above 150 or diastolic above 90 mm Hg)
3. Neurological conditions such as stroke, seizures, dementia or organic brain syndrome
4. Any condition likely to impair cognitive function such as mental retardation, attention deficit disorder or severe pharmacological sedation
5. Treatment for tobacco dependence in the last four months
6. Alcohol or substance abuse or dependence other than nicotine within the last 12 months
7. Pregnancy, verified by urine pregnancy test for females at first visit and in the beginning of each of the two patch administration sessions
8. Lactating

   Healthy controls, additional exclusion criterion:
9. Current psychiatric Axis I disorder or Axis II schizophrenia spectrum disorder, verified by Structured Clinical Interview for DSM-IV (SCID)

   Participants with mental illness, additional exclusion criterion:
10. Treated with benztropine (a nicotinic and muscarinic antagonist) or with an acetylcholine esterase inhibitor currently or within the last four weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2009-06-02; Study Completion 2013-06-11

PRIMARY OUTCOMES:
Cognitive task performance

SECONDARY OUTCOMES:
Measures of subjective state plasma concentrations of nicotine and metabolites genoytype with regards to genes that may affect nicotine response.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Adams CE, Stevens KE. Evidence for a role of nicotinic acetylcholine receptors in schizophrenia. Front Biosci. 2007 May 1;12:4755-72. doi: 10.2741/2424. PMID 17485411
- [Background] Apud JA, Weinberger DR. Treatment of cognitive deficits associated with schizophrenia: potential role of catechol-O-methyltransferase inhibitors. CNS Drugs. 2007;21(7):535-57. doi: 10.2165/00023210-200721070-00002. PMID 17579498
- [Background] Arinami T, Ishiguro H, Onaivi ES. Polymorphisms in genes involved in neurotransmission in relation to smoking. Eur J Pharmacol. 2000 Dec 27;410(2-3):215-226. doi: 10.1016/s0014-2999(00)00816-5. PMID 11134671